CLINICAL TRIAL: NCT01810497
Title: Analysis of the Influence of Different Protocols of Postoperative Elastic Bandage Use in the Results of Otoplasty
Brief Title: Analysis of Postoperative Bandage Use Protocols in Otoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Davi Reis Calderoni, Plastic Surgeon; Division of Plastic Surgery of the Faculty of Medical Sciences, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLASTICA-001
Record Dates: First submitted 2013-03-10; First posted 2013-03-13 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Prominent Ears
Keywords: External ear; Ear abnormalities; External ear cartilages

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seven-day bandage use (Active Comparator): Patients randomized and instructed to use of ear bandage 24h/day for seven days after otoplasty
  Interventions: Procedure: Use of ear bandage
- Thirty-day bandage use (Active Comparator): Patients randomized and instructed to use of ear bandage 24h/day for thirty days after otoplasty
  Interventions: Procedure: Use of ear bandage

INTERVENTIONS:
Procedure: Use of ear bandage — Elastic bandage to be used on the postoperative period of otoplasty, starting immediately after the procedure. To be used 24hours/day for the specified period.

SUMMARY:
The aim of the study is to investigate the possible influence of different durations of use of postoperative elastic bandaging (seven days vs. thirty days) in the results of otoplasty. We hypothesize that the duration of elastic bandage use has no significant influence on the incidence of relapse of prominence of the ears and need for reoperation.

ELIGIBILITY:
Inclusion Criteria:

* Congenital bilateral ear prominence
* 10 years-old or older
* No previous attempt of surgical treatment

Exclusion Criteria:

* Pregnant women
* Breastfeeding women
* Blod clotting disorders or current anticoagulant use
* Uncontrolled systemic diseases

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of re-operation | until 12 months

SECONDARY OUTCOMES:
Change from immediate postoperative period of helix-mastoid distance | 6 months
Change from immediate postoperative period of helix-mastoid distance | 12 months

OTHER OUTCOMES:
Incidence of hemorrhagic complications | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Davi R Calderoni, M.D., Principal Investigator — Division of Plastic Surgery, Faculty of Medical Sciences, University of Campinas - Unicamp
Locations (1):
- Unicamp Hospital, Campinas, São Paulo, Brazil